CLINICAL TRIAL: NCT06140732
Title: A Single-arm Phase 2 Study of Apatinib (Anti-PD-1) Combined With Camrelizumab (Anti-VEGFR ) in Patients With Advanced Chordoma
Brief Title: Apatinib Combined With Camrelizumab in Treating Participants With Advanced Chordoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XW-NS-ACCFC
Record Dates: First submitted 2023-11-08; First posted 2023-11-20 (Actual); Last update posted 2023-11-20 (Actual); Status verified 2023-10

CONDITIONS: Chordoma; Chemotherapy Effect
MeSH Terms: conditions — Chordoma | interventions — camrelizumab; apatinib

STUDY DESIGN:
Intervention Model Description: camrelizumab 200 mg iv/ q2w+ apatinib 375mg oral qd
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- camrelizumab combined with apatinib (Experimental): camrelizumab 200 mg iv/ q2w+ apatinib 375mg oral qd
  Interventions: Drug: camrelizumab and apatinib

INTERVENTIONS:
Drug: camrelizumab and apatinib — camrelizumab 200 mg iv/ q2w+ apatinib 375mg oral qd
  Other Names: Targeted therapy

SUMMARY:
This phase II trial studies how well Camrelizumab combined with Apatinib work in treating participants with chordoma that has spread to other places in the body, which may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the clinical benefit of the combination of Camrelizumab combined with Apatinib in patients with advanced chordomas by adverse events (AEs) and progression free survival (PFS).

SECONDARY OBJECTIVES:

I. Ascertain the safety of nivolumab in combination with relatlimab in subjects with metastatic or locally advanced/unresectable chordoma by the Overall survival (OS), objective response rate (MPR) and disease control rate (DCR)

EXPLORATORY OBJECTIVES:

I. Compare response rate (RR) and clinical benefit rate (CBR) in patients whose tumors are PD-L1+ and PD-L1- at baseline.

II. Compare RR and CBR in patients whose tumors are VEGFR+ and VEGFR- at baseline.

III. In the patients who are PD-L1 positive, compare RR and CBR in patients with 1% and 5% tumor membrane staining.

III. Determine the response to treatment based on the baseline mutation load. IV. Determine the ORR and CBR via Choi criteria.

OUTLINE:

To evaluate the safety and tolerability of carrilizol combined with apatinib in patients with recurrent, unresectable, chemotherapy-failed chordoma

After completion of study treatment, participants are followed up within 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 16 years old, male or female; 2. The physical status score of the Eastern Cancer Collaboration Group (ECOG) was 0-1; 3. Expected survival ≥3 months; 4. Patients with advanced chordoma confirmed by histopathology; 5. Imaging was available to evaluate the lesions. According to the evaluation criteria for solid tumor efficacy (RECIST 1.1, see Annex 2), there was at least one single-diameter measurable lesion, whose longest diameter was measured by spiral CT ≥ 10 mm; 6. All acute toxicities resulting from prior antitumor therapy were resolved to grade 0-1 (according to NCI CTCAE version 5.03) or to the level specified in the enrollment/exclusion criteria prior to enrollment (except for toxicities such as alopecia that the investigator determined did not pose a safety risk to the subject); If subjects undergo major surgery, they must have fully recovered from complications before starting treatment; 7. If the major organs function normally, the following criteria are met:

1. The standard of blood routine examination should be met (no blood transfusion and blood products within 14 days, no G-CSF and other hematopoietic stimulating factors are used to correct) :

   1. Hemoglobin (Hb) ≥ 80 g/L;
   2. Neutrophil count (ANC) ≥ 1.5×109/L;
   3. Platelet count (PLT) ≥ 80×109/L;
2. Biochemical examination shall meet the following standards:

   1. Total bilirubin (TBIL) < 1.5 ULN;
   2. ALT and AST < 2.5ULN, and < 5ULN in patients with liver metastasis; Alkaline phosphatase < 5ULN;
   3. Serum Cr ≤ ULN or endogenous creatinine clearance > 45 ml/min. 8. Women of childbearing age must have used reliable contraception or had a pregnancy test (serum or urine) within 7 days prior to enrol, with a negative result, and be willing to use an appropriate method of contraception during the trial period and 60 days after the last dose of the test drug. For men, consent to use appropriate methods of contraception or surgical sterilization during the trial period and for 120 days after the last dose of the trial drug; 9. The subjects voluntarily joined the study and signed the informed consent, with good compliance and follow-up.

Exclusion Criteria:

1. Except for those subjects whose toxicity had not recovered from previous antitumor therapy (concurrent chemoradiotherapy, surgical treatment) (alopecia, alkaline phosphatase, glutamine detranspeptase (GGT)) or who could be enrolled after discussion with the investigator and sponsor
2. Use of immunosuppressive drugs within 14 days prior to first use of carrilizumab, excluding nasal and inhaled corticosteroids or systemic steroid hormones at physiological doses (i.e., no more than 10 mg/ day of prednisolone or other corticosteroids at pharmacologically equivalent doses);
3. Previous treatment with anti-PD-1, anti-PD-L1, anti-VEGFR antibodies or anti-PD-L2 drugs or drugs that target another stimulus or synergistically inhibit T cell receptors (e.g., CTLA-4, OX-40, CD137);
4. Uncontrolled hypertension (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 90 mmHg, despite systematic medication);
5. Severe cardiovascular disease: Grade II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTc interval ≥450 ms for men and ≥470 ms for women); Grade Ⅲ to Ⅳ cardiac insufficiency (according to the New York Heart Society NYHA classification, see Annex 3), or left ventricular ejection fraction (LVEF) < 50% indicated by cardiac color ultrasound;
6. Patients with any active autoimmune disease or history of autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism) are not included;
7. The subjects were treated with bronchodilators and other systemic treatments, but their asthma control was unsatisfactory and they could not be included (those whose asthma had been completely relieved in childhood could be included without any intervention after adulthood).
8. Urine routine suggests urinary protein ≥ ++, or confirms 24-hour urinary protein volume ≥1.0g;
9. Abnormal coagulation function (INR >1.5 ULN or prothrombin time (PT) > ULN+4 seconds or APTT >1.5 ULN), have a tendency to bleed or are receiving thrombolytic or anticoagulant therapy; Note: Under the premise of INR ≤ 1.5, the use of low dose heparin (adult daily dose of 0.6 thousand to 12 thousand U) or low dose aspirin (daily dose of 100 mg or less) is permitted for preventive purposes;
10. A severe infection occurring within 4 weeks prior to the first dose (e.g., requiring intravenous antibiotic, antifungal, or antiviral medication), or an unexplained fever >38.5°C during the screening period/prior to the first dose;
11. Severe arteriovenous thrombosis events, such as cerebrovascular accidents (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, occurred within 12 months before enrollment;
12. Had undergone major surgery or severe traumatic injury, fracture or ulcer within 4 weeks prior to enrollment;
13. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active tuberculosis, active hepatitis B (HBV DNA ≥ 500 IU/ml), hepatitis C (hepatitis C antibody positive, And HCV-RNA is higher than the lower limit of detection method) or co-infected with hepatitis B and hepatitis C;
14. Patients with a clear history of allergy may have an underlying allergy or intolerance to the biologics of Apatinib and carrilizumab;
15. There are significant factors affecting the absorption of oral drugs, such as inability to swallow, chronic diarrhoea and intestinal obstruction. Or have cavity or perforation of viscera or sinus within 6 months;
16. Those who have a history of psychotropic drug abuse and cannot quit or have mental disorders;
17. Increases the risks associated with study participation or study drugs and, in the investigator's judgment, may result in other conditions for which the patient is not eligible for study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness: Progression-free survival (PFS) | 6 months
  To assess the clinical benefit of the combination of Camrelizumab combined with Apatinib in patients with advanced chordomas by adverse event and Progression-free survival.
Incidence and severity of AE | From date of start treatment until date of first documented of progression of withdrawal (through study completion, an average of 1 year).
  To assess the clinical benefit of the combination of Camrelizumab combined with Apatinib in patients with advanced chordomas by adverse event and Progression-free survival.

SECONDARY OUTCOMES:
Overall survival (OS), , disease | From date of start treatment until date of first documented of progression of withdrawal (through study completion, an average of 1 year).
  To assess the clinical benefit of the combination of Camrelizumab combined with Apatinib in patients with advanced chordomas by Overall survival (OS).
Objective response rate (OPR) | From date of start treatment until date of first documented of progression of withdrawal (through study completion, an average of 1 year).
  To assess the clinical benefit of the combination of Camrelizumab combined with Apatinib in patients with advanced chordomas by objective response rate (OPR)
Control rate (DCR) | From date of start treatment until date of first documented of progression of withdrawal (through study completion, an average of 1 year).
  To assess the clinical benefit of the combination of Camrelizumab combined with Apatinib in patients with advanced chordomas by disease control rate (DCR).

CONTACTS AND LOCATIONS:
Overall Officials: Zan Chen, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- BEIJING, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Somaiah N, Conley AP, Parra ER, Lin H, Amini B, Solis Soto L, Salazar R, Barreto C, Chen H, Gite S, Haymaker C, Nassif EF, Bernatchez C, Mitra A, Livingston JA, Ravi V, Araujo DM, Benjamin R, Patel S, Zarzour MA, Sabir S, Lazar AJ, Wang WL, Daw NC, Zhou X, Roland CL, Cooper ZA, Rodriguez-Canales J, Futreal A, Soria JC, Wistuba II, Hwu P. Durvalumab plus tremelimumab in advanced or metastatic soft tissue and bone sarcomas: a single-centre phase 2 trial. Lancet Oncol. 2022 Sep;23(9):1156-1166. doi: 10.1016/S1470-2045(22)00392-8. Epub 2022 Aug 4. PMID 35934010
- [Background] Liu C, Jia Q, Wei H, Yang X, Liu T, Zhao J, Ling Y, Wang C, Yu H, Li Z, Jiao J, Wu Z, Yang C, Xiao J. Apatinib in patients with advanced chordoma: a single-arm, single-centre, phase 2 study. Lancet Oncol. 2020 Sep;21(9):1244-1252. doi: 10.1016/S1470-2045(20)30466-6. PMID 32888455
- [Background] Chen Y, Jia Y, Liu Q, Shen Y, Zhu H, Dong X, Huang J, Lu J, Yin Q. Myocarditis related to immune checkpoint inhibitors treatment: two case reports and literature review. Ann Palliat Med. 2021 Jul;10(7):8512-8517. doi: 10.21037/apm-20-2620. Epub 2021 Jul 1. PMID 34263614
- [Background] Ulici V, Hart J. Chordoma. Arch Pathol Lab Med. 2022 Mar 1;146(3):386-395. doi: 10.5858/arpa.2020-0258-RA. PMID 34319396
- [Background] DeMaria PJ, Lee-Wisdom K, Donahue RN, Madan RA, Karzai F, Schwab A, Palena C, Jochems C, Floudas C, Strauss J, Marte JL, Redman JM, Dombi E, Widemann B, Korchin B, Adams T, Pico-Navarro C, Heery C, Schlom J, Gulley JL, Bilusic M. Phase 1 open-label trial of intravenous administration of MVA-BN-brachyury-TRICOM vaccine in patients with advanced cancer. J Immunother Cancer. 2021 Sep;9(9):e003238. doi: 10.1136/jitc-2021-003238. PMID 34479925
- [Result] Blay JY, Chevret S, Le Cesne A, Brahmi M, Penel N, Cousin S, Bertucci F, Bompas E, Ryckewaert T, Soibinet P, Boudou-Rouquette P, Saada Bouzid E, Soulie P, Valentin T, Lotz JP, Tosi D, Neviere Z, Cancel M, Ray-Coquard I, Gambotti L, Legrand F, Lamrani-Ghaouti A, Simon C, Even C, Massard C. Pembrolizumab in patients with rare and ultra-rare sarcomas (AcSe Pembrolizumab): analysis of a subgroup from a non-randomised, open-label, phase 2, basket trial. Lancet Oncol. 2023 Aug;24(8):892-902. doi: 10.1016/S1470-2045(23)00282-6. Epub 2023 Jul 7. PMID 37429302